CLINICAL TRIAL: NCT00627536
Title: A Double-Blind, Placebo-Controlled, Randomised Dose-Ranging Trial to Investigate the Efficacy of Avotermin (Juvista) in the Improvement of Scar Appearance When Applied to Approximated Wound Margins in Healthy Volunteers
Brief Title: Scar-Improvement Efficacy and Safety of a Single Intradermal Injection of Avotermin (Juvista) Administered Following Full-Thickness Skin Incisions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Mr Mark Cooper, Senior Vice President of Clinical Operations, Renovo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1001-0050
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2008-03

CONDITIONS: Cicatrix
Keywords: scarring, Juvista, avotermin, transforming growth factor beta 3, TGFB3
MeSH Terms: conditions — Cicatrix; Arrhythmogenic Right Ventricular Dysplasia, Familial, 1 | interventions — TGFB3 protein, human; Transforming Growth Factor beta3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Experimental): Avotermin 5ng/100μL/linear cm wound margin
  Interventions: Drug: Avotermin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 3 (Experimental): Avotermin 50ng/100μL/linear cm wound margin
  Interventions: Drug: Avotermin
- 4 (Placebo Comparator): Placebo matched to avotermin 50ng/100μL/linear cm
  Interventions: Drug: Placebo
- 5 (Experimental): Avotermin 200ng/100μL/linear cm
  Interventions: Drug: Avotermin
- 6 (Placebo Comparator): Placebo matched to avotermin 200ng/100μL/linear cm
  Interventions: Drug: Placebo
- 7 (Experimental): Avotermin 500ng/100μL/linear cm wound margin
  Interventions: Drug: Avotermin
- 8 (Placebo Comparator): Placebo matched to avotermin 500ng/100μL/linear cm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avotermin — A single intradermal injection of avotermin administered at the dose to both margins of a full-thickness incision immediately following closure.
  Other Names: Juvista, RN1001, transforming growth factor beta 3
  Arms: 1; 3; 5; 7
Drug: Placebo — Matched to avotermin dosage strength
  Other Names: None applicable
  Arms: 2; 4; 6; 8

SUMMARY:
This study was undertaken to investigate the scar-improvement efficacy and safety of a single dose of avotermin (Juvista) injection into skin incisions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-85 years who had given written informed consent.
* Subjects with a body mass index within 15 to 35 kg/m2.
* Subjects with clinically acceptable results for the laboratory tests
* Female subjects of child bearing potential who are using acceptable method(s) of contraception.

Exclusion Criteria:

* Subjects with history or evidence of hypertrophic or keloid scarring.
* Subjects with tattoos or previous scars within 3cm of the area to be incised.
* Subjects with prior surgery in the area to be incised within one year of the first dosing day.
* Subjects with a history of a bleeding disorder; receiving anti-coagulant or anti-platelet therapy.
* Subjects with evidence of any past or present clinically significant disease that may affect the endpoints of the trial.
* Subjects with a clinically significant skin disorder that is chronic or currently active.
* Subjects with any clinically significant medical condition or history that would impair wound healing.
* Subjects with a history of drug hypersensitivity to any of the drugs or dressings used in this trial.
* Subjects who are taking, or have taken any investigational product or participated in a clinical trial in the three months prior to first trial dose administration.
* Subjects who are taking regular, continuous, oral corticosteroid therapy.
* Subjects undergoing investigations or changes in management for an existing medical condition.
* Subjects with a history of drug abuse, or with a positive drugs of abuse test for cocaine, amphetamines, metamphetamines, opiates or benzodiazepines during the screening period.
* Subjects who are considered unlikely to complete the trial for whatever reason.
* Subjects with a clinically significant neurological impairment or disease.
* Subjects with any active infection.
* Subjects who are pregnant or lactating.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Scar appearance | 7 months

SECONDARY OUTCOMES:
Safety: adverse events, local tolerability | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: James Bush, MBChB, Principal Investigator — Renovo
Locations (1):
- Renovo Clinical Trials Unit, Manchester, United Kingdom